CLINICAL TRIAL: NCT05765149
Title: Sleep Trajectories Among Pregnant Women and Its Impact on Maternal and Infant Outcomes: a Prospective Cohort Study
Brief Title: A Cohort Study on Sleep Disorders During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20220305-R
Record Dates: First submitted 2023-02-02; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hair samples will be collected before delivery and 3 months after delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleep Cohort: This is an observational study. We plan to recruit 1000 pregnant women during 10-13 weeks gestational age to build a sleep cohort. Their sleep changes during pregnancy will be recorded for identifying similar groups.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study, no intervention will be implemented.

SUMMARY:
The goal of this observational study is to: 1) determine the prevalence of sleep disorders in pregnancy and the early postpartum; 2) identify factors associated with sleep disturbance during pregnancy and the early postpartum; 3) describe the progression of sleep quality and quantity as gestational age; 4) determine if sleep is associated with adverse perinatal outcomes. Participants were asked to wear a forehead sleep recorder for 4 consecutive days and to complete a sleep questionnaire at ten timepoints: at 3 months, 4 months, 5 months, 6 months, 7 months, 8 months, and 9 months pregnant and at 1 month, 2 months and 3 months postpartum.

DETAILED DESCRIPTION:
There is a high incidence of sleep disturbances globally, especially among pregnant women. Long-term sleep disorders seriously affect the quality life of individuals, and it becomes undoubtedly an important public health problem. Studies have shown that sleep disorders during pregnancy can have short-term and long-term adverse effects on both mothers and their babies. In addition, sleep during pregnancy exhibits different characteristics at different stages. Most of the existing studies are based on the overall development trend to study sleep characteristics, ignoring potential individual differences. Based on the concept of precision medicine, this study intends to establish a cohort focusing on the sleep health of pregnant women, and carry out continuous home sleep monitoring of pregnant women from both subjective and objective perspectives. The aim of this study is, firstly, to explore the longitudinal change characteristics, potential classification and influencing factors of sleep during pregnancy; secondly, to analyze the differences in maternal and infant adverse outcomes among pregnant women with different sleep development trajectories. The final goal is to reveal the exposure window of maternal and infant adverse outcomes caused by sleep, thus improving the accuracy of outcome prediction, and promoting the development of accurate and personalized sleep management programs.

ELIGIBILITY:
Inclusion Criteria:

1. Gestation age ≤ 13 weeks + 6 days
2. 20 years old ≤ Age ≤ 40 years old
3. Singleton pregnancy
4. Give informed consent and able to participated

Exclusion Criteria:

1. Unmarried, divorced or widowed
2. Women who suffered severe physical or mental illness
3. Women who suffered death, abortion, stillbirth or neonatal death during the study
4. Women who are participating in other studies
5. Other reasons

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is mainly from maternal hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Preterm birth | delivery
  Preterm birth refers to a body born before 37 weeks of gestation. It will be identified according to the medical history records.
Caesarean section | delivery
  Caesarean section refers to a baby delivered through an incision in the mother's abdomen. It will be identified according to the medical history records.
Postpartum depression symptoms at 1 month after delivery | 1 month after delivery
  Postpartum depression symptoms at 1 month after delivery will be measured by the Edinburgh postpartum depression scale (EPDS).
Postpartum depression symptoms at 2 months after delivery | 2 months after delivery
  Postpartum depression symptoms at 2 months after delivery will be measured by the Edinburgh postpartum depression scale (EPDS).
Postpartum depression symptoms at 3 months after delivery | 3 months after delivery
  Postpartum depression symptoms at 3 months after delivery will be measured by the Edinburgh postpartum depression scale (EPDS).

SECONDARY OUTCOMES:
1-minute Apgar score | 1 minute after delivey
  Apgar is a quick test performed on a baby at 1 and 5 minutes after birth. It will be identified according to the medical history records.
5-minute Apgar score | 5 minutes after delivey
  Apgar is a quick test performed on a baby at 1 and 5 minutes after birth. It will be identified according to the medical history records.
Infant's length | delivey
  It will be identified according to the medical history records.
Infant's weight | delivey
  It will be identified according to the medical history records.

CONTACTS AND LOCATIONS:
Overall Officials: Man Wang, Master, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No